CLINICAL TRIAL: NCT07277140
Title: Impact of Iron Deficiency With and Without Anemia on Arrhythmic Events and Resting ECG Abnormalities in Patients Hospitalized With Heart Failure
Brief Title: Impact of Iron Deficiency on Arrhythmic Events and Resting ECG Abnormalities in Patients Hospitalized With Heart Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Mohamed Sadek, Cardiology Resident, Principal Investigator, Assiut University
Other Study IDs: Iron deficiency& Heart failure
Record Dates: First submitted 2025-09-23; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Iron Deficiency
MeSH Terms: conditions — Heart Failure; Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The relationship between iron deficiency (with or without anemia) and arrhythmic risk or ECG abnormalities in hospitalized HF patients remains poorly characterized. This is particularly relevant in settings where advanced iron therapies (e.g., intravenous iron supplementation) may not be readily available, and where simple clinical and electrocardiographic markers could help identify high-risk patients by evaluating the impact of iron deficiency (with and without anemia) arrhythmic events and resting ECG changes among patients admitted with heart failure. Understanding these associations may offer insights into the arrhythmogenic potential of iron deficiency and support the integration of iron status assessment into routine risk stratification and management of HF patients.

DETAILED DESCRIPTION:
Heart failure (HF) is a major global health problem, associated with high morbidity, mortality, and frequent hospitalizations. Beyond impaired cardiac function, HF is recognized as a systemic syndrome involving a wide range of metabolic, inflammatory, and hematologic disturbances that contribute to disease progression and adverse outcomes. Iron deficiency has emerged as a prevalent and clinically relevant comorbidity, affecting up to 55% of chronic HF patients and in up to 80% of those with AHF, even in the absence of overt anemia.

Iron plays a central role in cellular energy metabolism, oxidative phosphorylation, and mitochondrial function, processes that are especially critical in the metabolically demanding environment of the myocardium.

In patients with HF, anemia and iron deficiency has been associated with reduced exercise capacity, impaired quality of life, and increased risk of hospitalization, cardiovascular and all-cause mortality. While the impact of iron deficiency on functional status and survival has been widely investigated, its potential influence on cardiac electrical activity remains less well studied.

Emerging evidence suggests that iron deficiency may contribute to electrophysiological instability by promoting oxidative stress, altering repolarization, and impairing myocardial conduction. This could create a potential substrate for arrhythmias, which are a major cause of morbidity in patients with HF. Moreover, subtle resting electrocardiographic (ECG) abnormalities, such as QT prolongation, T-wave changes, or conduction delays, may reflect early electrical remodeling in the context of iron deficiency-even in the absence of clinically apparent arrhythmias

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years) admitted to Assiut University Heart Hospital with a clinical diagnosis of heart failure (new-onset or decompensated).

Includes all ejection fraction categories (HFrEF, HFmrEF, and HFpEF).

Availability of 12-lead ECG, serum iron studies (ferritin, transferrin saturation, serum iron), and routine laboratory tests.

Willingness to participate and provide informed consent.

Exclusion Criteria:

Known history of primary electrical disorders (e.g., Brugada syndrome, Long QT syndrome, etc.).

Recent intravenous iron therapy or blood transfusion within the past 3 months.

End-stage renal disease requiring dialysis.

Known anemia due to non-iron-deficiency causes (e.g., hemolytic anemia, active malignancy, etc.).

Severe electrolyte imbalances (e.g., significant hypo-/hyperkalemia, hypo-/hypermagnesemia).

Active systemic infection, chronic inflammatory conditions, or recent chemotherapy.

severe valvular lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) admitted with heart failure over a period of one year at Assiut University Heart Hospital (AUHH)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of anemia and iron deficiency in hospitalized patients with HF | through study completion, an average of 1 year
  The proportion of patients admitted with heart failure who are found to have anemia and/or iron deficiency during hospitalization. Anemia is defined according to WHO criteria (Hb <13 g/dL in men, <12 g/dL in women). Iron deficiency is defined as ferritin <100 ng/mL, or ferritin 100-299 ng/mL with transferrin saturation <20%.
Incidence of arrhythmic events in hospitalized HF patients with and without iron deficiency possible | through study completion, an average of 1 year
  The proportion of hospitalized heart failure patients who experience arrhythmic events (such as atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or clinically significant bradyarrhythmias) during admission. Patients will be categorized based on the presence or absence of iron deficiency (defined by ferritin <100 ng/mL, or ferritin 100-299 ng/mL with transferrin saturation <20%).

SECONDARY OUTCOMES:
Resting ECG abnormalities in hospitalized HF patients with and without iron deficiency | through study completion, an average of 1 year
  The prevalence and types of resting ECG abnormalities (e.g., atrial fibrillation/flutter, QRS prolongation >120 ms, ST-T changes, pathological Q waves, left ventricular hypertrophy, bundle branch blocks, premature ventricular complexes) in hospitalized heart failure patients. Patients will be stratified according to the presence or absence of iron deficiency (defined as ferritin <100 ng/mL, or ferritin 100-299 ng/mL with transferrin saturation <20%).
Correlation between iron parameters, anemia status, and resting electrophysiologic parameters on 12-lead ECG | through study completion, an average of 1 year
  This outcome evaluates the correlation between iron status indicators (serum ferritin, transferrin saturation, and serum iron levels) and anemia-defined according to WHO criteria (hemoglobin <13 g/dL in men, <12 g/dL in women)-with resting electrophysiologic parameters obtained from a standard 12-lead ECG.
  Each electrophysiologic parameter will be correlated separately with continuous iron and hemoglobin values
Association between iron parameters (and anemia) and electrophysiologic parameters | through study completion, an average of 1 year
  Assessment of the relationship between iron status (ferritin, transferrin saturation, serum iron) and anemia (defined by WHO criteria: Hb <13 g/dL in men, <12 g/dL in women) with resting electrophysiologic parameters on 12-lead ECG. Parameters include:
  Rhythm: sinus rhythm, atrial fibrillation/flutter, ventricular arrhythmias
  Conduction: PR interval, QRS duration, bundle branch block
  Repolarization: QT/QTc interval, ST-T abnormalities
  Heart rate variability (if available)
  Patients will be stratified according to presence/absence of iron deficiency and anemia, and correlations will be examined between continuous iron parameters and ECG metrics.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Crespo-Leiro MG, Anker SD, Maggioni AP, Coats AJ, Filippatos G, Ruschitzka F, Ferrari R, Piepoli MF, Delgado Jimenez JF, Metra M, Fonseca C, Hradec J, Amir O, Logeart D, Dahlstrom U, Merkely B, Drozdz J, Goncalvesova E, Hassanein M, Chioncel O, Lainscak M, Seferovic PM, Tousoulis D, Kavoliuniene A, Fruhwald F, Fazlibegovic E, Temizhan A, Gatzov P, Erglis A, Laroche C, Mebazaa A; Heart Failure Association (HFA) of the European Society of Cardiology (ESC). European Society of Cardiology Heart Failure Long-Term Registry (ESC-HF-LT): 1-year follow-up outcomes and differences across regions. Eur J Heart Fail. 2016 Jun;18(6):613-25. doi: 10.1002/ejhf.566. PMID 27324686
- [Result] Salah HM, Minhas AMK, Khan MS, Pandey A, Michos ED, Mentz RJ, Fudim M. Causes of hospitalization in the USA between 2005 and 2018. Eur Heart J Open. 2021 Jun 15;1(1):oeab001. doi: 10.1093/ehjopen/oeab001. eCollection 2021 Aug. PMID 35919090
- [Result] Boulet J, Sridhar VS, Bouabdallaoui N, Tardif JC, White M. Inflammation in heart failure: pathophysiology and therapeutic strategies. Inflamm Res. 2024 May;73(5):709-723. doi: 10.1007/s00011-023-01845-6. Epub 2024 Mar 28. PMID 38546848
- [Result] McDonagh T, Damy T, Doehner W, Lam CSP, Sindone A, van der Meer P, Cohen-Solal A, Kindermann I, Manito N, Pfister O, Pohjantahti-Maaroos H, Taylor J, Comin-Colet J. Screening, diagnosis and treatment of iron deficiency in chronic heart failure: putting the 2016 European Society of Cardiology heart failure guidelines into clinical practice. Eur J Heart Fail. 2018 Dec;20(12):1664-1672. doi: 10.1002/ejhf.1305. Epub 2018 Oct 12. PMID 30311713
- [Result] Pantopoulos K, Porwal SK, Tartakoff A, Devireddy L. Mechanisms of mammalian iron homeostasis. Biochemistry. 2012 Jul 24;51(29):5705-24. doi: 10.1021/bi300752r. Epub 2012 Jul 9. PMID 22703180
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL. Corrigendum to: 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Oct 21;42(40):4194. doi: 10.1093/eurheartj/ehab648. No abstract available. PMID 34520521
- [Result] Chung YJ, Luo A, Park KC, Loonat AA, Lakhal-Littleton S, Robbins PA, Swietach P. Iron-deficiency anemia reduces cardiac contraction by downregulating RyR2 channels and suppressing SERCA pump activity. JCI Insight. 2019 Apr 4;4(7):e125618. doi: 10.1172/jci.insight.125618. eCollection 2019 Apr 4. PMID 30779710